CLINICAL TRIAL: NCT06589609
Title: A Phase 1 Study of FluBHPVE6E7 Immunotherapy in Patients With HPV16- Associated Oropharyngeal Squamous Cell Carcinoma
Brief Title: Phase 1 Clinical Trial of FluBHPVE6E7 Immunotherapy for HPV16-Associated Oropharyngeal Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: BlueSky Immunotherapies GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BS-03; 2024-514413-36-00 (EU CTIS Number)
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Oropharyngeal Squamous Cell Carcinoma (SCC)
Keywords: immunotherapy; Oropharyngal squamous cell carcinoma; HPV-16; Human papilloma virus; cancer; Head and neck cancer
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Neoplasms; Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): FlubHPVE6E7
  Interventions: Biological: FluBHPVE6E7

INTERVENTIONS:
Biological: FluBHPVE6E7 — Intratumoral administration for first dose followed by intramuscular administration for subsequent doses at recommended dose level and determined schedule.

SUMMARY:
A clinical study of an immunotherapy in patients with head or neck cancers associated with the HPV16 virus

DETAILED DESCRIPTION:
Squamous cell carcinomas of the head and neck (HNSCC) rank as the sixth most common cancer globally, with approximately 575,000 new cases diagnosed each year. In recent years, there has been a rising incidence in younger patients who have limited exposure to traditional risk factors such as smoking and alcohol. This increase is closely associated with HPV infection, particularly HPV-16, which is strongly linked to oropharyngeal cancer. Treatment for HPV-positive oropharyngeal squamous cell carcinoma (OPSCC) is highly individualized, depending on the disease stage, patient comorbidities, and personal preferences. In this phase 1 study, patients with HPV-16-associated OPSCC are being treated with the immunotherapeutic delNS-vector expressing the HPV-16 oncogenes E6 and E7, administered both intratumorally and intramuscularly.

ELIGIBILITY:
Inclusion criteria:

* Female or male patients, 18-65 years of age, with newly diagnosed, histologically confirmed p16- and HPV16-positive oropharyngeal squamous cell carcinoma with locoregional advanced disease including the following stages:

  * T2N2-3, M0
  * T3N0-3, M0
  * T4N0-3, M0
* Primary tumour accessible for biopsy and intratumoural administration
* No evidence of distant metastatic disease (HPV16-positive secondary tumours are permissible)
* Karnofsky 100 - 70 (ECOG 0 or 1)
* Life expectancy of at least 6 months
* Normal screening ECG or screening ECG with no clinically significant findings requiring immediate treatment, as judged by the investigator
* Women of childbearing potential: Negative serum pregnancy test at screening
* Agree to use a reliable form of contraception until the end of the study treatment period.
* Provides written informed consent

Exclusion criteria:

* Distant metastases
* Secondary, not HPV16-associated, malignancy
* History of malignancy other than the target malignancy to be investigated in this trial unless a complete remission was achieved at least 2 years prior to study entry AND no additional therapy is required during the study period
* Clinically significant out of range haematological, renal or hepatic laboratory tests which cannot be explained by the underlying disease
* Any vaccination within 1 week before day 0
* Active significant viral infections including influenza, CMV, and EBV within 4 weeks before receiving study treatment
* Co-infection with hepatitis B, hepatitis C, or HIV or having other immune deficient states
* Influenza-like illness (ILI) within 4 weeks before day 0
* Known hypersensitivity to Tamiflu or any of its components
* Pregnancy, breastfeeding
* Serious, concomitant disorder, including active systemic infection requiring treatment
* Proven or suspected systemic lupus erythematosus, thyroiditis, inflammatory bowel disease including Crohn's disease or multiple sclerosis
* Immunosuppression including any concurrent condition requiring the continued use of systemic steroids, or the use of immunosuppressive agents, disease modifying doses of anti-rheumatic drugs (e.g., azathioprine, cyclophosphamide, cyclosporine, methotrexate), and biologic disease modifying drugs such as TNF-α inhibitors (e.g. infliximab, adalimumab or etanercept). Corticosteroids must be discontinued > 4 weeks prior to day 0 of study medication administration. Eye drops or ear drops containing corticosteroids are permissible.
* Prior major surgery within 4 weeks before day 0
* Any current significant cardiac, hepatic or renal disease or history of clinically significant, medically unstable disease (e.g. chronic renal failure; angina, myocardial ischemia or infarction, congestive heart failure, cardiomyopathy, or clinically significant arrhythmias)
* Participation in another experimental protocol/use of investigational drug within two months before day 0
* Any condition that, in the judgment of the investigator, might prevent safe participation in the study or interfere with study objectives
* Unability to comply with the protocol requirements

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-08-23 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
Frequency and severity of adverse events (AEs) | 7 days
  To assess the severity of the adverse event is assessed according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 5.0.

SECONDARY OUTCOMES:
Intralesional T-cell infiltration | 24 weeks
  To assess the intralesional T-cell infiltration in tumour tissue available from surgery or biopsy by immunohistological staining.
Biodistribution | 24 weeks
  To evaluate the presence of FluBHPVE6E7 by quantification of FluBHPVE6E7 genome copies in nasal secretion samples by RT-qPCR (copies per ml blood).
Virus recovery in oropharyngeal secretion samples | 7 days
  To evaluate the presence of FluBHPVE6E7 by quantification of FluBHPVE6E7 genome copies in oropharyngeal secretion samples by RT-qPCR (copies per sample).
Virus recovery in saliva | 7 days
  To evaluate the presence of FluBHPVE6E7 by quantification of FluBHPVE6E7 genome copies in saliva samples by RT-qPCR (copies per sample).
Frequency and severity of adverse events (AEs) | 24 weeks
  To assess the severity of the adverse event according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 5.0.
Disease-free survival (DFS) | 60 months
  To assess the length of time after treatment during which the patient remains free from any signs or symptoms of the disease.
Overall survival (OS) | 60 months
  To assess the length of time from the start of treatment or diagnosis until the death of the patient from any cause.
Induction of HPV-specific T-cell response following FluBHPVE6E7 administration | 24 weeks
  To assess the induction of HPV16 E6- and E7-specific T-cells (%) by IFN-gamma ELISPOT analysis.
Hemagglutination Inhibition (HAI) Geometric Mean Titers (GMTs) following FluBHPVE6E7 administration | 24 weeks
  To assess the induction of systemic vector-specific antibodies by HAI assay.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No